CLINICAL TRIAL: NCT04870359
Title: Pre-emptive Increase of Immunosuppressive Treatments in Lupus Nephritis Patients With Asymptomatic Serological Reactivation
Brief Title: Pre-emptive Treatments in Lupus Nephritis Patients With Serological Reactivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: United Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW-16-074
Record Dates: First submitted 2017-07-03; First posted 2021-05-03 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-emptive Treatment (Prednisolone and/or AZA/MMF) (Active Comparator): 1. Increase prednisolone to 0.4-0.5 mg/kg/day; taper by 5 mg every 2 weeks to reach 15mg/day; then further reduce by 2.5 mg every 2 week and aim to reach 5-7.5 mg/day after 12 weeks.
  2. Adjustment of the 2nd agent would be as follows:
     1. For patients who receive AZA <75mg/day; increase the dose of AZA to 75 mg/day.
     2. For patients who receive MMF <1g/day, increase the dose of MMF to 1g/day.
  Interventions: Procedure: Pre-emptive increase of immunosuppressive treatments; Drug: Prednisolone and/or AZA/MMF
- Control (No Intervention): Current immunosuppressive regimen and dosage should remain unchanged until the development of renal or extra-renal flares which required increase/change in immunosuppression.

INTERVENTIONS:
Procedure: Pre-emptive increase of immunosuppressive treatments — 1. Increase prednisolone to 0.4-0.5 mg/kg/day; taper by 5 mg every 2 weeks to reach 15mg/day; then further reduce by 2.5 mg every 2 week and aim to reach 5-7.5 mg/day after 12 weeks.
  2. Adjustment of the 2nd agent would be as follows:
     1. For patients who receive AZA <75mg/day; increase the dose of AZA to 75 mg/day.
     2. For patients who receive MMF <1g/day, increase the dose of MMF to 1g/day.
  Arms: Pre-emptive Treatment (Prednisolone and/or AZA/MMF)
Drug: Prednisolone and/or AZA/MMF — Prednisolone and/or AZA/MMF
  Arms: Pre-emptive Treatment (Prednisolone and/or AZA/MMF)

SUMMARY:
The optimal management of asymptomatic serological reactivation (ASR) in lupus nephritis (LN) patients remained undefined. This project aims to investigate the impact of pre-emptive treatment on disease relapse in LN patients who experienced ASR.

DETAILED DESCRIPTION:
LN patients who presented with ASR [defined as 1) increase in anti-dsDNA >100 IU/mL , with or without drop in serum complement; or 2) increase in anti-dsDNA to higher than the normal range and >2 times of the preceding value, with or without drop in serum complement; and 3) Absence of renal or systemic manifestations of SLE) will be randomized to receive pre-emptive increase in immunosuppression or had their current immunosuppressive therapies unchanged.

Patients will be followed at 4-, 12-, 24-wk and then every 12 weeks up to 24 months to monitor for renal or extra-renal relapses. Bloods and urine will be collected for measurement of renal and serological parameters, and also B cell signatures.

Primary outcomes: Renal Flare (denoted as proteinuria >1g/D; presence of urinary RBC >30 hpf/RBC casts, or increase in SCr >15% and positive anti-dsDNA)

Secondary outcomes:

* Safety & tolerability of pre-emptive increase of immunosuppressive treatments
* Extra-renal flares
* Renal function at 24 months
* Changes in serological parameters

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven lupus nephritis who experienced an episode of Asymptomatic Serological Flare (ASF) as defined by:

  1. Increase in anti-dsDNA to >100 IU/mL, with or without drop in serum complement levels OR
  2. Increase in anti-dsDNA to higher than the normal range and more than two times of the preceding value, with or without drop in serum complement levels

     AND
  3. Absence of renal or systemic manifestation of SLE.

Exclusion Criteria:

1. Patients who cannot provide informed consent.
2. Patients whom the clinicians opined to have excessively high risk of infection or malignancy.
3. Patients who are pregnant or lactating.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-04-21 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Renal Flare | Within 24 months
  A composite endpoint denoted by proteinuria >1g/day, presence of urinary RBC >30/hpf or RBC casts, or increase in serum creatinine by 15% compared with baseline, and anti-DNA antibody titre above the upper limit of normal

SECONDARY OUTCOMES:
Infections requiring hospitalization | 24 months
Extra-renal flares | 24 months
Serum creatinine levels | 24 months
Changes in anti-dsDNA | 24 months
Changes in C3 | 24 months
Changes in Hba1c | 24 months
Changes in fasting glucose | 24 months
Changes in LDL levels | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Desmond YH Yap, MBBS (HK). MD (HK), Principal Investigator — Queen Mary Hospital, The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong, Hong Kong
  - United Christian Hospital, Hong Kong